CLINICAL TRIAL: NCT01257477
Title: Research Study to Evaluate LOTRONEX® in Severe IBS-D: Analysis of Current Clinical Practice Environment
Brief Title: LOTRONEX® in Severe Diarrhea-Predominant Irritable Bowel Syndrome (IBS-D)
Acronym: RELIANCE
Status: Completed | Type: Observational
Sponsor: Prometheus Laboratories (Industry)
Responsible Party: Sponsor
Other Study IDs: 10LOT01
Record Dates: First submitted 2010-12-07; First posted 2010-12-09 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: Diarrhea; IBS; Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
An observational study to evaluate LOTRONEX® in women with severe IBS-D in the current clinical practice setting.

DETAILED DESCRIPTION:
This observational study will evaluate the effect of Lotronex® as used in the current clinical practice setting on symptom relief, specifically, improvement in bowel habits and IBS pain. Patients planning to initiate commercially available LOTRONEX® therapy will be consented for study participation. Patients will complete study questionnaires related to bowel symptoms, prior therapies, quality of life, productivity loss and treatment outcome. Investigators will also be asked to complete questionnaires related to the patient's disease characteristics, patient progress on study medication and treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Be a female between 18 and 65 years of age (inclusive) at Visit 1.
2. Sign and date a written informed consent form prior to the initiation of any study-related activities, including discontinuation of any prohibited medications.
3. Be diagnosed with severe, diarrhea-predominant IBS.
4. Have experienced chronic IBS symptoms lasting 6 months or longer.
5. Have not responded adequately to other IBS therapy.
6. Be able to read, understand and sign the informed consent and, if applicable, an Authorization to Use and Disclose Protected Health Information form (consistent with Health Insurance Portability and Accountability Act of 1996 [HIPAA] legislation), answer the study questionnaires, communicate with the investigator, and understand and comply with protocol requirements.

Exclusion Criteria:

1. Has had a period of 3 consecutive days without a bowel movement in the past 14 days.
2. In the past 14 days, has had evidence of chronic or severe constipation, or has a history of chronic or severe constipation, or a history of sequelae from constipation.
3. Has recurrent bowel obstruction of the small intestine or colon.
4. Has had bloody diarrhea or abdominal pain with rectal bleeding in the past 14 days (except rectal bleeding due to hemorrhoids).
5. Has a known biochemical or anatomical abnormality of the gastrointestinal tract.
6. Has a history of thrombophlebitis or hypercoagulable state.
7. Has a history of atherosclerosis.
8. Has any medical or surgical condition that in the judgment of the investigator makes the patient an inappropriate candidate for Lotronex® therapy (e.g., an unstable cardiovascular, autoimmune, renal, hepatic, pulmonary, endocrine, metabolic, gastrointestinal, hematologic, or neurological condition; recent or ongoing malignancy; evidence of hepatic dysfunction; or renal impairment.)
9. Mental impairment of inability to understand the medication guide and instructions for study participation or refusal to comply with protocol.
10. Current (within 7 days from start of Lotronex® use) use of fluvoxamine.
11. Chronic (≥ 6 months) use of narcotics or opioids.
12. The patient has used an investigational drug or participated in an investigational study within 30 days of Visit 1/ Screening Visit.
13. The patient is hypersensitive or has a known negative response to 5-HT3 antagonists.
14. Had a significant adverse event during previous treatment with Lotronex® or is currently using Lotronex®.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women ≥ 18 years of age with severe diarrhea-predominant IBS, who have chronic IBS symptoms lasting 6 months or longer and who have not responded adequately to other IBS therapy will be eligible to enroll in the study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2010-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in stool consistency | At Week 4 and Week 12
  Stool consistency as measured by the Bristol Stool Form Scale. Change from baseline at Weeks 4 and 12 will be determined.
IBS pain severity | At Weeks 4 and 12
  Pain intensity as measured by the 11-point numeric rating scale (NRS) will be averaged for each 4-week interval. Change from baseline at Weeks 4 and 12 will be determined.

SECONDARY OUTCOMES:
Change from baseline in quality of life scores (IBSQOL). | Week 12
  Change from baseline in IBSQOL scores will be calculated at Week 12.
Change from baseline stool frequency. | Week 4 and Week 12
  Stool frequency will be measured as the mean number of times per day that stools were passed, and will be averaged for each 4-week interval. Change from baseline at Weeks 4 and 12 will be determined
Change from baseline in fecal urgency. | Week 4 and Week 12
  Proportion of days with fecal urgency will be calculated for each 4-week interval and change from baseline will be determined at 4 and 12 weeks.
Change from baseline in lost productivity. | 12 Weeks
  Lost workplace productivity and number of days IBS symptoms interfered with social/leisure and household activities will be determined at baseline and week 12. Change from baseline to week 12 will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Emil Chuang, MD, Study Director — Prometheus Therapeutics and Diagnostics
Locations (67):
- United States (67):
  - Gastroenterology Consultants Inc., Tuscaloosa, Alabama
  - Digestive Health Research Unit, Scottsdale, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Adam D. Karns, MD, Beverly Hills, California
  - Behavioral Research Specialists, LLC, Irvine, California
  - Torrance Clinical Research, Lomita, California
  - Community Clinical Trials, Orange, California
  - Inland Gastroenterology Medical Associates, Redlands, California
  - Digestive Care Associates, San Carlos, California
  - Clinical Applications Laboratories, Inc., San Diego, California
  - Precision Research Institute, LLC, San Diego, California
  - Delta Waves Sleep Disorders & Research Center, Colorado Springs, Colorado
  - Clinical Research of the Rockies, Lafayette, Colorado
  - Gastroenterology Associates of Fairfield County, Bridgeport, Connecticut
  - Consultants for Clinical Research of South Florida, Boynton Beach, Florida
  - Sanitas Research, Coral Gables, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Southern Clinical Research Consultants, Hollywood, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Advanced Gastroenterology Associates, LLC, Palm Harbor, Florida
  - Gulf Regions Clinical Research Institute, Pensacola, Florida
  - Accord Clinical Research, LLC, Port Orange, Florida
  - Bearss Medical, Tampa, Florida
  - Florida Medical Clinic, PA, Zephyrhills, Florida
  - Illinois Gastroenterology Group, LLC/Northwest Gastroenterologists, Arlington Heights, Illinois
  - GI Solutions, Chicago, Illinois
  - Investigative Clinical Research of Indiana, LLC, Elwood, Indiana
  - Gastrointestinal Clinic of Quad Cities, Davenport, Iowa
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Metropolitan Gastroenterology Group, PC, Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Commonwealth Clinical Studies, Brockton, Massachusetts
  - Troy Gastroenterology, PC, Troy, Michigan
  - Gastroenterology Associates of Western Michigan, Wyoming, Michigan
  - Center for Digestive and Liver Diseases, Inc., Mexico, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Howard Guss, DO, Ocean City, New Jersey
  - Synergy First, LLC, Brooklyn, New York
  - Long Island Clinical Research Associates, Great Neck, New York
  - New York Center for Clinical Research, Lake Success, New York
  - Concorde Medical Group, New York, New York
  - NY Center for Women's Health Research, New York, New York
  - Asheville Gastroenterology Associates, PA, Asheville, North Carolina
  - Carolina Digestive Diseases, Greenville, North Carolina
  - Carolinas Research Associates, Harrisburg, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Consultants for Clinical Research of Cincinnati, Cincinnati, Ohio
  - Gastroenterology Research Consultants of Greater Cincinnati, Cincinnati, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - Gastroenterology United of Tulsa, Tulsa, Oklahoma
  - The Orgeon Clinic - West Hills Gastroenterology, Portland, Oregon
  - Pennsylvania Research Institute, Bensalem, Pennsylvania
  - Research Across America, Reading, Pennsylvania
  - Anderson Gastroenterology Associates, LLC, Anderson, South Carolina
  - Franklin Gastroenterology, PLLC, Franklin, Tennessee
  - HCCA Clinical Research Solutions, Jackson, Tennessee
  - Murfreesboro Medical Clinic, Murfreesboro, Tennessee
  - Academy of Clinical Research, Arlington, Texas
  - ARAYVAN Clinical Research, Arlington, Texas
  - Austin Center for Clinical Research, Austin, Texas
  - Trinity Clinical Research, Carrollton, Texas
  - Digestive Health Center, Pasadena, Texas
  - Spring Gastroenterology, Spring, Texas
  - Granger Medical Clinic, West Valley City, Utah
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Advanced Gastroenterology, Vancouver, Washington

REFERENCES:
- [Derived] Lacy BE, Nicandro JP, Chuang E, Earnest DL. Alosetron use in clinical practice: significant improvement in irritable bowel syndrome symptoms evaluated using the US Food and Drug Administration composite endpoint. Therap Adv Gastroenterol. 2018 May 8;11:1756284818771674. doi: 10.1177/1756284818771674. eCollection 2018. PMID 29774051